CLINICAL TRIAL: NCT04759495
Title: Comparison of CGM in Non-randomised Real Life Study of Real-time and Intermittently Scanned Systems in Patients With Type 1 Diabetes
Brief Title: Is Real-time CGM Superior to Flash Glucose Monitoring in Real Life Study (CORRIDA LIFE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Soupal, MD, Principal Investigator, Charles University, Czech Republic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CORRIDA LIFE
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Continuous Glucose Monitoring; Flash Glucose Monitoring; Hypoglycaemia; Time in Range
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- rtCGM (Experimental): Patients with use of the DEXCOM G5 or G6 system (real time continuous glucose monitoring).
  Interventions: Device: Continuous Glucose Monitoring Dexcom G5 and G6 system (real-time continuous glucose monitoring)
- FGM (Experimental): Patients with use of the FreeStyle Libre Flash system (flash glucose monitoring).
  Interventions: Device: Continuous Glucose Monitoring FreeStyle Libre Flash system (flash glucose monitoring)

INTERVENTIONS:
Device: Continuous Glucose Monitoring Dexcom G5 and G6 system (real-time continuous glucose monitoring) — rtCGM is used in Type 1 diabetic patients to improve glucose control and to minimize or avoid severe hypoglycaemia.
  Arms: rtCGM
Device: Continuous Glucose Monitoring FreeStyle Libre Flash system (flash glucose monitoring) — FGM is used in Type 1 diabetic patients to improve glucose control and to minimize or avoid severe hypoglycaemia.
  Arms: FGM

SUMMARY:
The aim of the investigator's study is to compare real-time continuous glucose monitoring (rt-CGM) and flash glucose monitoring (FGM) in adult patients with Type 1 Diabetes (T1D) in real life practice during 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients with T1D naive to rt-CGM and FGM
* Type 1 diabetes for > 1 year
* ≥ 18 years old
* CSII without automatic functions or MDI

Exclusion Criteria:

* previous rtCGM or FGM use
* treatment with insulin pump with automatic functions
* severe noncompliance
* known severe diabetic retinopathy and/or macular edema
* lactation, pregnancy, or intending to become pregnant during the study
* a condition likely to require MRI
* use of acetaminophen-containing medication
* unwillingness to use the study device for >70% of time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in glycated haemoglobin (HbA1c) | Up to 13 months
  Differences between HbA1c values in the Run in period and after 12 month of follow-up and differences of HbA1c between groups.

SECONDARY OUTCOMES:
Percentage of time in hypoglycemic ranges | Up to 13 months
  <3.9 mmol/L [70 mg/dl] and <3.0 mmol/L [54 mg/dl]
Percentage of time in target ranges | Up to 13 months
  3.9-10.0 mmol/L [70-180 mg/dl]
Percentage of time in hyperglycemic ranges | Up to 13 months
  >10.0 mmol/L [180 mg/dl] and >13.9 mmol/L [250 mg/dl]
Changes in glycemic variability | Up to 13 months
  Expressed as the standard deviation
Mean sensor glucose concentration | Up to 13 months
  Measured by rtCGM or FGM
Incidence of severe hypoglycaemia | Up to 13 months
  Requiring third-party assistance to treat
Incidence of severe ketoacidosis | Up to 13 months
  Requiring hospitalization
Incidence of skin reaction, infection or hematoma at the site of insertion of the sensor | Up to 13 months
  Skin reaction, infection or hematoma reported by patients

CONTACTS AND LOCATIONS:
Overall Officials: Jan Soupal, Principal Investigator — Charles University, Prague
Locations (1):
- 3rd Department of Internal Medicine, 1st Faculty of Medicine, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haskova A, Radovnicka L, Petruzelkova L, Parkin CG, Grunberger G, Horova E, Navratilova V, Kade O, Matoulek M, Prazny M, Soupal J. Real-time CGM Is Superior to Flash Glucose Monitoring for Glucose Control in Type 1 Diabetes: The CORRIDA Randomized Controlled Trial. Diabetes Care. 2020 Nov;43(11):2744-2750. doi: 10.2337/dc20-0112. Epub 2020 Aug 28. PMID 32859607
- [Background] Fullerton B, Jeitler K, Seitz M, Horvath K, Berghold A, Siebenhofer A. Intensive glucose control versus conventional glucose control for type 1 diabetes mellitus. Cochrane Database Syst Rev. 2014 Feb 14;2014(2):CD009122. doi: 10.1002/14651858.CD009122.pub2. PMID 24526393
- [Background] Soupal J, Petruzelkova L, Flekac M, Pelcl T, Matoulek M, Dankova M, Skrha J, Svacina S, Prazny M. Comparison of Different Treatment Modalities for Type 1 Diabetes, Including Sensor-Augmented Insulin Regimens, in 52 Weeks of Follow-Up: A COMISAIR Study. Diabetes Technol Ther. 2016 Sep;18(9):532-8. doi: 10.1089/dia.2016.0171. Epub 2016 Aug 2. PMID 27482825
- [Background] Soupal J, Petruzelkova L, Grunberger G, Haskova A, Flekac M, Matoulek M, Mikes O, Pelcl T, Skrha J Jr, Horova E, Skrha J, Parkin CG, Svacina S, Prazny M. Glycemic Outcomes in Adults With T1D Are Impacted More by Continuous Glucose Monitoring Than by Insulin Delivery Method: 3 Years of Follow-Up From the COMISAIR Study. Diabetes Care. 2020 Jan;43(1):37-43. doi: 10.2337/dc19-0888. Epub 2019 Sep 17. PMID 31530663
- [Background] Beck RW, Riddlesworth T, Ruedy K, Ahmann A, Bergenstal R, Haller S, Kollman C, Kruger D, McGill JB, Polonsky W, Toschi E, Wolpert H, Price D; DIAMOND Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Adults With Type 1 Diabetes Using Insulin Injections: The DIAMOND Randomized Clinical Trial. JAMA. 2017 Jan 24;317(4):371-378. doi: 10.1001/jama.2016.19975. PMID 28118453
- [Background] Oskarsson P, Antuna R, Geelhoed-Duijvestijn P, Krӧger J, Weitgasser R, Bolinder J. Impact of flash glucose monitoring on hypoglycaemia in adults with type 1 diabetes managed with multiple daily injection therapy: a pre-specified subgroup analysis of the IMPACT randomised controlled trial. Diabetologia. 2018 Mar;61(3):539-550. doi: 10.1007/s00125-017-4527-5. Epub 2017 Dec 23. PMID 29273897
- [Background] Bolinder J, Antuna R, Geelhoed-Duijvestijn P, Kroger J, Weitgasser R. Novel glucose-sensing technology and hypoglycaemia in type 1 diabetes: a multicentre, non-masked, randomised controlled trial. Lancet. 2016 Nov 5;388(10057):2254-2263. doi: 10.1016/S0140-6736(16)31535-5. Epub 2016 Sep 12. PMID 27634581
- [Background] Heinemann L, Freckmann G, Ehrmann D, Faber-Heinemann G, Guerra S, Waldenmaier D, Hermanns N. Real-time continuous glucose monitoring in adults with type 1 diabetes and impaired hypoglycaemia awareness or severe hypoglycaemia treated with multiple daily insulin injections (HypoDE): a multicentre, randomised controlled trial. Lancet. 2018 Apr 7;391(10128):1367-1377. doi: 10.1016/S0140-6736(18)30297-6. Epub 2018 Feb 16. PMID 29459019
- [Derived] Radovnicka L, Haskova A, Do QD, Horova E, Navratilova V, Mikes O, Cihlar D, Parkin CG, Grunberger G, Prazny M, Soupal J. Lower Glycated Hemoglobin with Real-Time Continuous Glucose Monitoring Than with Intermittently Scanned Continuous Glucose Monitoring After 1 Year: The CORRIDA LIFE Study. Diabetes Technol Ther. 2022 Dec;24(12):859-867. doi: 10.1089/dia.2022.0152. Epub 2022 Sep 22. PMID 36037056